CLINICAL TRIAL: NCT00608010
Title: Day 3 Embryo Cryopreservation: Metabolic and Viability Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Basak Balaban, Chief Embryologist, American Hospital of Istanbul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AH-ART-06/13
Record Dates: First submitted 2008-01-22; First posted 2008-02-06 (Estimated); Last update posted 2008-02-06 (Estimated); Status verified 2008-01

CONDITIONS: Fertilization in Vitro; Preservation of Supernumerary Embryos
Keywords: Preservation of supernumerary embryos in an IVF program
MeSH Terms: interventions — Vitrification

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Vitrification
  Interventions: Procedure: Vitrification
- 2 (Active Comparator): Slow freezing
  Interventions: Procedure: Slow freezing

INTERVENTIONS:
Procedure: Vitrification — Embryos were vitrified according to a previously described technique
  Arms: 1
Procedure: Slow freezing — Embryos were frozen with slow freezing technique
  Arms: 2

SUMMARY:
Embryo preservation through freezing plays a significant role in human assisted reproduction. It provides an opportunity for patients to have more than one attempt following an ovarian stimulation cycle, thereby decreasing the exposure of patients to exogenous gonadotrophins and improving cumulative pregnancy rates. The purpose of this study is to compare effectiveness of two different freezing methods.

ELIGIBILITY:
Inclusion Criteria:

* ICSI with own gametes
* Couples who did not wish to cryopreserve their excess embryos for possible transfer in a future cyle
* Donating excess embryos for research purposes

Exclusion Criteria:

* Embryos derived from surgically retrieved spermatozoa
* Blastocysts
* Embryos of low quality (Grade 3 or 4 according to Hardarson)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2006-10; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Blastocyst development rate | 3 days after thawing

CONTACTS AND LOCATIONS:
Overall Officials: Basak Balaban, BSc, Principal Investigator — American Hospital of Istanbul
Locations (1):
- American Hospital of Istanbul, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Balaban B, Urman B, Ata B, Isiklar A, Larman MG, Hamilton R, Gardner DK. A randomized controlled study of human Day 3 embryo cryopreservation by slow freezing or vitrification: vitrification is associated with higher survival, metabolism and blastocyst formation. Hum Reprod. 2008 Sep;23(9):1976-82. doi: 10.1093/humrep/den222. Epub 2008 Jun 10. PMID 18544577